CLINICAL TRIAL: NCT01432275
Title: Ease of Use of New Blood Glucose Meter With In-built Insulin Calculator at Home Study
Acronym: IHUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ADC-PMS-INX-11011
Record Dates: First submitted 2011-09-09; First posted 2011-09-12 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; SMBG; Insulin calculator
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADC, Then Comparator, Then ADC With Calculator (Experimental): Subject used the ADC blood glucose meter for 7 days with the insulin calculator not activated, followed by a comparator blood glucose meter for 7 days. For the last 10 days the subject used the ADC blood glucose meter with insulin calculator active.
  Interventions: Device: ADC blood glucose meter; Device: Comparator blood glucose meter; Device: ADC blood glucose meter with insulin calculator active
- Comparator, Then ADC, Then ADC With Calculator (Experimental): Subject used a comparator blood glucose meter for 7 days, followed by the ADC blood glucose meter for 7 days, with the insulin calculator not activated. For the last 10 days the subject used the ADC blood glucose meter with insulin calculator active.
  Interventions: Device: ADC blood glucose meter; Device: Comparator blood glucose meter; Device: ADC blood glucose meter with insulin calculator active

INTERVENTIONS:
Device: ADC blood glucose meter — Subjects used the FreeStyle InsuLinx with the insulin calculator not activated. Subjects had not previously used the FreeStyle InsuLinx meter.
  Other Names: Abbott Freestyle InsuLinx
Device: Comparator blood glucose meter — Subjects were randomly assigned one of the comparator meters. Subjects had not previously used the assigned comparator meter.
  Other Names: Roche Accu-Chek Aviva Nano; Lifescan Verio Pro or; Bayer Contour USB
Device: ADC blood glucose meter with insulin calculator active — Subjects used the FreeStyle InsuLinx with the insulin calculator activated.
  Other Names: Abbott FreeStyle InsuLinx

SUMMARY:
The aim of this study is to evaluate user preference and ease of use of the FreeStyle InsuLinx system, compared to current methodology, when used at home by subjects with diabetes.

Subjects will also be comparing the ease of use of the FreeStyle InsuLinx system with comparator meters.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 or 2 diabetes on a bolus regime (U100 insulin), one or more bolus injections per day for at least 6 months;
* Age 18 yrs and above;
* Regularly testing SMBG 3 or more times per day;
* Willingness to test at least 4 times per day.

Exclusion Criteria:

* Know to require a bolus injection of more than 50U in a single dose;
* Has previously used either the InsuLinx or assigned comparison meter;
* Participated in structured diabetes management training in the last 6 months
* Is currently on an insulin pump;
* Has concomitant disease that, in the Investigator's opinion, may compromise patient safety;
* Is participating in another study of a glucose monitoring device or drug that could affect glucose measurements or glucose management;
* Female subject who is pregnant or planning to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shenaz Ramtoola, Principal Investigator — Royal Blackburn Hospital
Locations (7):
- United Kingdom (7):
  - Tameside Hospital NHS Foundation Trust, Ashton-under-Lyne
  - Ayr Hospital, Ayr
  - Royal United Hospital, Bath
  - Royal Blackburn Hospital, Blackburn
  - North Manchester Diabetes Centre, Crumpsall
  - Ipswich Hospital NHS Trust, Ipswich
  - Greenwood & Sneinton Family Medical Centre, Nottingham

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 179 subjects were enrolled on this study, 164 completed the study.
Pre-assignment Details: One subject was excluded due to not meeting all inclusion criteria, one subject withdrew before randomisation.
Period: First BG Meter System (7 Days)
Arm/Group | ADC, Then Comparator, Then ADC With Calculator | Comparator, Then ADC, Then ADC With Calculator
Started | 90 | 87
Completed | 90 | 84
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Second BG Meter System (7 Days)
Arm/Group | ADC, Then Comparator, Then ADC With Calculator | Comparator, Then ADC, Then ADC With Calculator
Started | 90 | 84
Completed | 88 | 81
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: ADC With Calculator (10 Days)
Arm/Group | ADC, Then Comparator, Then ADC With Calculator | Comparator, Then ADC, Then ADC With Calculator
Started | 88 | 81
Completed | 85 | 79
Not Completed | 3 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Per Protocol Population: Subjects who completed the study.
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 145
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81
  Male | 83
Region of Enrollment [Number; unit: participants]
  United Kingdom | 164
Type of Diabetes [Number; unit: participants]
  Type 1 | 128
  Type 2 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall User Preference for the FreeStyle InsuLinx System Compared to Current Method.
Description: Overall user preference of the FreeStyle InsuLinx system as a diabetes management tool when compared against their usual method.
Time Frame: 25 days
Population: A comparator blood glucose meter was used for 7 days and a FreeStyle InsuLinx for 7 days (insulin calculator inactive). For the last 10 days a FreeStyle InsuLinx with the insulin calculator activated was used. Each subject was assigned one of the three competitor systems. Subjects had not previously used any study systems. Analysis per protocol.
Measure: Number; unit: participants
Groups:
- Per Protocol Population: Subjects completing the study using the FreeStyle InsuLinx Blood Glucose Meter and one of the comparator blood glucose meters
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 164
participants | 125
Statistical Analysis 1: Comparison: Per Protocol Population; Test type: Superiority or Other; p < 0.0001, Binomial test; Comparison to 27 participants that preferred their usual method to FreeStyle InsuLinx. Twelve(12) participants did not have a preference

2. Secondary Outcome: Preference Questionnaire (Insulin Calculator Not Activated)
Description: Result for the question: "The meter the subject would change to"
Time Frame: 25 days (results recorded after the two 7 day periods)
Population: Subjects used a comparator blood glucose meter for 7 days and a FreeStyle InsuLinx meter for 7 days (insulin calculator deactivated). Subjects then completed a preference questionnaire. Each subject was assigned one of the three competitor systems. Subjects had not previously used either study device. Analysis per protocol.
Measure: Number; unit: participants
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 164
participants
  Subject would change to FreeStyle InsuLinx | 98
  Subject would change to a comparison meter | 32
  Not likely to change / not sure / missing answer | 34

ADVERSE EVENTS:
Time Frame: Adverse events collected from enrolment to completion by last subject (up to 2 months).
Groups:
- ADC Blood Glucose Meter: ADC blood glucose meter for 7 days with the insulin calculator not activated.
- Comparator Blood Glucose Meter: Comparator blood glucose meter for 7 days.
- ADC Blood Glucose Meter With Calculator: ADC blood glucose meter for 10 days with the insulin calculator active.
Arm/Group | ADC Blood Glucose Meter | Comparator Blood Glucose Meter | ADC Blood Glucose Meter With Calculator
Serious Adverse Events (participants affected / at risk) | 2/177 | 0/177 | 1/169
Other Adverse Events (participants affected / at risk) | 0/178 | 0/178 | 0/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADC Blood Glucose Meter (N=177) | Comparator Blood Glucose Meter (N=177) | ADC Blood Glucose Meter With Calculator (N=169)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Admitted with severe abdominal pain following hysterectomy
Hypoglycaemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) — Hypoglycaemia leading to seizure, not related to study or device.
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Vomiting - admitted to hospital for less than 24 hrs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days